CLINICAL TRIAL: NCT03436992
Title: Estrogen-Mediated Impairments of Vascular Health in Diabetes
Brief Title: Estrogen and Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ryan Harris, Associate Professor, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2 and D; 1R01HL137087-01A1 (NIH)
Record Dates: First submitted 2018-02-13; First posted 2018-02-19 (Actual); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Estrogen, Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Women with type 1 diabetes (Experimental): Women with type 1 diabetes will be randomly assigned to 1 of the 3 interventions (Antioxidant cocktail, Resveratrol, or placebo)
  Interventions: Dietary Supplement: Antioxidant Cocktail; Dietary Supplement: Resveratrol; Other: Placebo
- Healthy control women (No Intervention): Healthy women who participate will receive no intervention and serve as controls.
- Men with type 1 diabetes (Experimental): Men with type 1 diabetes will be randomly assigned to 1 of the 3 interventions (AOX cocktail, Resveratrol, or placebo)
  Interventions: Dietary Supplement: Antioxidant Cocktail; Dietary Supplement: Resveratrol; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Antioxidant Cocktail — Vitamin C, Vitamin E, alpha lipoic acid
  Arms: Men with type 1 diabetes; Women with type 1 diabetes
Dietary Supplement: Resveratrol — 1500 mg trans-resveratrol
  Arms: Men with type 1 diabetes; Women with type 1 diabetes
Other: Placebo — placebo
  Arms: Men with type 1 diabetes; Women with type 1 diabetes

SUMMARY:
Diabetes has recently been referred to as "the epidemic of the 21st century". The reason why women with type 1 diabetes have a 2-3 fold greater risk of cardiovascular disease (CVD) compared to men with type 1 diabetes is unknown.The purpose of this study is to investigate whether or not estrogen contributes to vascular dysfunction in premenopausal women with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Both men and premenopausal
* Normal menstrual cycle interval of 25-35 days for at least 3 previous cycles
* All races
* Clinical diagnosis of insulin-dependent type 1 diabetes (patients only)

Exclusion Criteria:

* Clinical diagnosis of hepatic, cardiovascular, or renal disease
* Uncontrolled Diabetes (HbA1c>9%)
* Diabetic complications (i.e. macrovascular, microvascular, or autonomic)
* Proteinuria
* Uncontrolled Hypertension (>140/90 mmHg on therapy)
* Hormonal use of birth control (past 3 months)
* Pregnancy
* Oligomenorrhea
* Direct vasoactive medications (i.e. nitrates)
* Anti-estrogens (i.e. SERMs)
* Plycystic ovarian syndrome (defined by NIH guidelines-hyperandrogenic anovulation)
* Undetectable Anti-Mullerian Hormone (AMH) following screening

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 143 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Harris, PhD, CES, Principal Investigator — Augusta University
Locations (2):
- United States (2):
  - Augusta University, Augusta, Georgia
  - Georgia Prevention Institute, Augusta, Georgia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: These results were based on a subset (n=57) of the total enrollment of 143.
Groups:
- T1M Women: women with type 1 diabetes
- Controls: apparently healthy women
Period: Overall Study
Arm/Group | T1M Women | Controls
Started | 32 | 25
Completed | 32 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T1M Women | Controls | Total
Number analyzed (Participants) | 32 | 25 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (6) | 24 (6) | 25 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 25 | 57
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 11 | 20
  White | 23 | 14 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 163.5 (7.0) | 165.4 (5.8) | 164.3 (6.5)
Weight [Mean (Standard Deviation); unit: kg] | 72.8 (17.6) | 68.4 (15.8) | 70.9 (16.8)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.2 (5.7) | 24.5 (4.7) | 26.0 (5.4)
MAP [Mean (Standard Deviation); unit: mm Hg] | 87 (8) | 83 (7) | 85 (8)
CRP [Mean (Standard Deviation); unit: mg/L] — C-Reactive Protein
  mg/L | 5.4 (8.3) | 1.2 (1.3) | 3.6 (6.6)
TC [Mean (Standard Deviation); unit: mg/dL] — Total Cholesterol
  mg/dL | 178 (41) | 163 (35) | 171 (39)
HDL [Mean (Standard Deviation); unit: mg/dL] | 58 (17) | 53 (13) | 56 (15)
LDL [Mean (Standard Deviation); unit: mg/dL] | 98 (42) | 88 (39) | 94 (41)
TRIG [Mean (Standard Deviation); unit: mg/dL] — Triglycerides
  mg/dL | 76 (45) | 63 (28) | 70 (39)
TC/HDL ratio [Mean (Standard Deviation); unit: ratio] | 3.2 (1.1) | 3.2 (0.8) | 3.2 (1.0)
HbA1c [Mean (Standard Deviation); unit: percent] | 8.6 (1.7) | 5.2 (0.3) | 7.1 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: FMD/Shear
Description: Flow-Mediated Dilation (FMD) controlled for shear
Time Frame: ~ 2 weeks. Acquired at Menses and Late Follicular phase.
Measure: Mean (Standard Deviation); unit: %/s^-1
Arm/Group | T1M Women | Controls
Number analyzed (Participants) | 32 | 25
%/s^-1
  Menses | 0.182 (0.068) | 0.206 (0.100)
  Late Follicular | 0.155 (0.059) | 0.219 (0.110)

ADVERSE EVENTS:
Time Frame: Baseline to Post testing (~2 weeks)
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | T1M Women | Controls
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/25
Other Adverse Events (participants affected / at risk) | 0/32 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT03436992/Prot_SAP_000.pdf